CLINICAL TRIAL: NCT01419613
Title: Motivational Interviewing to Promote Physical Activity in Breast Cancer Survivors
Brief Title: Promoting a Healthier Lifestyle Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-16265
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: healthy lifestyle; physical activity; behavior; motivational; interview; breast cancer survivor
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Behavior | interventions — Motivational Interviewing; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing (Experimental)
  Interventions: Behavioral: Motivational Interviewing
- Physical Activity Counseling (Active Comparator)
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Motivational Interviewing — Breast cancer survivors will receive general information on how to adopt healthy lifestyle behaviors.
  Arms: Motivational Interviewing
Behavioral: Counseling — The control group of breast cancer survivors will receive counseling on how to increase their level of physical activity.
  Arms: Physical Activity Counseling

SUMMARY:
The purpose of this study is to find out if a counseling program the investigators have developed can help breast cancer survivors adopt a healthier lifestyle.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of two groups. One group of breast cancer survivors will receive general information on how to adopt healthy lifestyle behaviors. The other group of breast cancer survivors will receive counseling on how to increase their level of physical activity.

Participants will have three consultations with a health counselor. The first two consultations will take place in-person and the third consultation will take place via telephone. Participants will also be asked to complete questionnaires assessing their physical and mental well-being, their dietary habits, and their physical activity habits at four time-points: in-person during their first study visit, via mail or through an online survey 6 weeks later, in-person 12 weeks later, and via mail or through an online survey 24 weeks later. Additionally, during their first study visit and 12 weeks later, their level of aerobic fitness will be tested by having participants walk a long hallway for six minutes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age;
* be capable of speaking and reading English;
* be diagnosed with stage 0-II breast cancer;
* be currently disease free;
* have been treated surgically for breast cancer;
* have completed chemotherapy and/or radiotherapy at least three months but no more than two years prior;
* be physically able to exercise as measured by the Physical Activity Readiness Questionnaire-Revised (Thomas, Reading, & Shephard, 1992) ;
* be currently physically inactive as measured by the Godin Leisure Time Exercise Questionnaire (Godin & Shepard, 1985); and
* be contemplating increasing physical activity as measured by the Exercise Stages of Change - Short Form (Marcus, Selby, Niaura, & Rossi, 1992).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Increased Activity After Motivational Interviewing | 24 Weeks Per Participant
  The primary objective of this study is to evaluate the efficacy of a brief Motivational Interviewing (MI) based intervention, relative to a time and attention control intervention (healthy lifestyle counseling), in promoting physical activity among early-stage breast cancer survivors who are physically inactive but are contemplating increasing their level of physical activity.

SECONDARY OUTCOMES:
Number of Participants With Desired Impact on Symptoms After Motivational Interviewing | 24 Weeks Per Participant
  The secondary objectives of this study are (1) to examine the impact of the MI intervention on depressive symptoms, fatigue, vigor, and aerobic fitness; and
Number of Participants With Desired Effects From Increased Physical Activity | 24 Weeks Per Participant
  (2) to explore whether the degree of change in physical activity acts as a mediator of the expected benefits of the MI intervention on depressive symptoms, fatigue, vigor, and aerobic fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B. Jacobsen, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States